CLINICAL TRIAL: NCT00792311
Title: Tsui Test as a Predictor of Bupivacaine Consumption in Labour Epidurals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose C.A. Carvalho, Mount Sinai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-02
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Pain
Keywords: Tsui test; Epidural Analgesia
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tsui test (Experimental): Tsui test administration.
  Interventions: Procedure: Tsui test

INTERVENTIONS:
Procedure: Tsui test — The stimulator is set at frequency of 1Hz with 200ms pulse width and the current output ranging from 0 to 20 mA. The current output will be carefully increased from zero until motor activity is detected up to a maximum of 20 mA.

SUMMARY:
Low current electrical stimulation test, also called the Tsui test, has been used successfully to confirm the catheter location in the epidural space in various patient populations. The results of this study will show whether or not doing a Tsui test can predict inadequate epidural analgesia early in the course of placing the epidural, so that the appropriate measures could be applied immediately upon gathering unfavorable results.

DETAILED DESCRIPTION:
Despite its very high success rate, the epidural technique remains a rather blind technique, and failures continue to occur. The incidence and reasons for failure are not well understood. The Tsui test is not routinely performed with each epidural catheter insertion, but rather it is used when there is suspicion about the catheter location.

In this study, the Tsui test will be performed twice during the epidural procedure, and bupivacaine consumption will be recorded for the first 2 hours.

Information gained from this study could have great impact in clinical practice, since the incidence of inadequate labor analgesia is still relatively high (10-20%), leading to maternal distress and disappointing labor experience.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age requesting an epidural for labor and delivery
* Cervix dilated 0-5 cm and pain VAS>6
* Able to communicate in English
* Informed consent

Exclusion Criteria:

* Refusal to provide written informed consent
* Patients unable to communicate in English
* Contraindication to regional anesthesia
* Allergy or hypersensitivity to lidocaine, bupivacaine or fentanyl
* Sedatives or opioids received prior to insertion of epidural catheter
* Abnormal vertebral anatomy, such as previous spine surgery and scoliosis
* Coexisting neurological disorders
* Patients with implanted electronic devices

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Consumption of bupivacaine in mg/hour in the first 2 hours of epidural anesthesia | 2 hours

SECONDARY OUTCOMES:
Incidence of inadequate epidural block. | 2 hours
Current (mA) needed to elicit motor response; 1. before test dose and 2. 5 minutes after test dose. | 5 minutes
Contraction pattern elicited by the Tsui test at baseline and after test dose. | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada